CLINICAL TRIAL: NCT05091684
Title: Administration of Fibrinogen Concentrate for Refractory Bleeding in Hematological Patients With Intensive Chemotherapy-induced Thrombocytopenia - Analysis Using Viscoelastic Haemostatic Assay (FORMAT)
Brief Title: Administration of Fibrinogen Concentrate for Refractory Bleeding
Acronym: FORMAT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Only one patient was included in this study due to overly restrictive inclusion and exclusion criteria.
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0201; 2021-000990-10 (EudraCT Number)
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Hematological Patients; Bleeding; Platelet Refractoriness
Keywords: hematology; intensive chemotherapy; platelet transfusion; thrombocytopenia; fibrinogen
MeSH Terms: conditions — Hemorrhage; Thrombocytopenia | interventions — Fibrinogen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibrinogen (Experimental): Patients with refractory thrombocytopenia, following intensive chemotherapy, and presenting grade ≥ 2 hemorrhagic symptoms, will receive adjuvant fibrinogen administration and platelet transfusions.
  Interventions: Drug: Fibrinogen Concentrate Human

INTERVENTIONS:
Drug: Fibrinogen Concentrate Human — Refractory transfused patients who present grade ≥ 2 hemorrhagic symptoms will receive a single injection of fibrinogen concentrate (1.5g) followed by platelet transfusion within 2 hours. Blood sampling will be done at different time points to measure clot viscoelasticity: at baseline, after fibrinogen injection, after platelet transfusion and the day after transfusion or before the next platelet transfusion if < 24 hours.

SUMMARY:
Platelet transfusions are widely employed to prevent or treat bleeding episodes in patients with thrombocytopenia. Patients with bone marrow failure secondary to haematological malignancy and chemotherapy frequently receive prophylactic platelet transfusion when platelet level reaches 10x109.L-1, to avoid spontaneous major bleeding. Due to immune or nonimmune factors, platelet refractoriness may be observed and is defined as a repeated suboptimal response to platelet transfusions with lower-than-expected post-transfusion count increments. The management of patients with alloimmunization is complex and prophylactic platelet support is no longer indicated. Therefore, platelet refractoriness remains a clinically challenging complication.

DETAILED DESCRIPTION:
To date, no specific therapeutic strategy has been proposed for platelet refractoriness, in cancer patients who are both at high risk of bleeding and thrombosis. Interestingly, fibrinogen is a critical hemostatic protein required for both prevention and treatment of bleeding as it provides a matrix and mesh network essential for clot formation, amplification and strength. Fibrinogen repletion, primarily with the use of fibrinogen concentrates for acquired bleeding, has been reported in clinical settings including surgery, trauma, and obstetrics. However, its use as adjuvant therapy for patients requiring massive transfusion is not yet a widely approved indication, especially in hematological patients. Therefore, the evidence regarding timing, efficacy and safety of fibrinogen administration in massively transfused hematological patients is scarce. This study aims at evaluating whether fibrinogen administration to transfused and refractory patients with on-going bleeding could affect the viscoelastic test of clotting function.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to a social security regimen or beneficiary of the same
* Signed written informed consent form
* Confirmed diagnosis of a hematological malignancy and undergoing intensive chemotherapy, autologous stem cell transplantation or allogeneic stem cell transplantation
* Grade ≥ II hemorrhagic symptoms according to WWorld Health Organization classification
* Failure or impossibility to use Human Leucocyte Antigen-matched platelet unit
* Body weight between 38 and 78 Kgs
* Transfusion refractoriness as defined by Corrected count increment ≤ 5 and platelet level < 20.109.L-1

Exclusion Criteria:

* Pregnant women
* Patient under guardianship or deprived of his liberty or any condition that may affect the patient's ability to understand and sign the informed consent
* Refusing participation
* Patient presenting non-malignant hematological disease
* Patient with high plasmatic concentration of fibrinogen (>5g/L)
* Patient who received fibrinogen within 20 days before inclusion
* Contra-indication to fibrinogen (fibrinogen concentrate) or any excipient (fibrinogen concentrate)
* Patient with disseminated intravascular coagulopathy
* Patient with thromboembolic history
* Patient who received L-Asparaginase or acquired hypofibrinogenemia following treatment by L-Asparaginase
* Patient with known risk of thrombophilia (deficiency for antithrombin 3, C protein or factor V)
* Patient with anti-thrombotic treatment (anti-platelet or anti-coagulant therapy) at the time of enrolment
* Elevated body temperature ≥ 38.5°C
* Hospital stay for invasive surgery
* Patient with acute myeloid leukemia during the induction phase of chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Maximal clot elasticity (viscoelastic test of clotting function) | 3 hours
  Measurement of viscoelastic test of clotting function represented by the maximal clot elasticity based on the maximal clot firmness from the EXTEM (EXtrinsically activated test) curve, between blood sampling before fibrinogen administration and blood sampling after platelet transfusion

SECONDARY OUTCOMES:
Comparison of viscoelastic test of clotting function before and after treatment using EXTEM (EXtrinsically activated test) and FIBTEM (fibrin clot obtained by platelet inhibition with cytochalasin D) curves (Fibrinogen) | 24 hours
  Measurement of viscoelastic test of clotting function to determine the contribution of fibrinogen in clotting (before fibrinogen, after fibrinogen, after fibrinogen + platelet transfusion)
Comparison of viscoelastic test of clotting function before and after treatment using EXTEM (EXtrinsically activated test) and FIBTEM (fibrin clot obtained by platelet inhibition with cytochalasin D) curves (platelets) | 24 hours
  Measurement of viscoelastic test of clotting function to determine the contribution of platelets in clotting (baseline, after fibrinogen + platelet transfusion)
Comparison of viscoelastic test of clotting function before and after treatment using EXTEM (EXtrinsically activated test) and FIBTEM (fibrin clot obtained by platelet inhibition with cytochalasin D) curves (platelets) | 24 hours
  Measurement of viscoelastic test of clotting function and comparison depending on platelet characteristics
Incidence of hemorrhagic and thrombotic events | 2 months
  Proportions of patients experiencing bleeding and thrombotic events
Incidence of adverse events | 2 months
  Proportions of patients experiencing adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Chalayer, MD, PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No